CLINICAL TRIAL: NCT00502697
Title: Tennessee Connections for Better Birth Outcomes
Acronym: BBO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Blue Cross Blue Shield (Other); Nurses for Newborns Foundation (Other)
Responsible Party: Principal Investigator, Melanie Lutenbacher, Associate Professor of Nursing and Medicine (General Pediatrics), Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 070684
Record Dates: First submitted 2007-07-16; First posted 2007-07-18 (Estimated); Results first posted 2016-03-16 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Preterm Birth
Keywords: preterm; prematurity; home visitation; system of care
MeSH Terms: conditions — Premature Birth | interventions — Postnatal Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Targeted Nurse Home Visits (Experimental): Advanced practice nurses provide targeted behavioral interventions during home visits. These visits were in addition to regularly scheduled conventional prenatal and postpartum clinic visits. Specific protocols guided nurse interventions related to tobacco use, substance use and misuse, stress management, dental health, maternal infections, perinatal depressive symptoms, family violence, reproductive life plans and continuity of care. Home visits were continued in the postpartum period (through 18 months post-delivery) with a continued focus on risk factors identified during the prenatal period and internatal health care.
  Interventions: Behavioral: Targeted Nurse Home Visits; Other: Conventional prenatal/postpartum care
- Conventional prenatal/postpartum care (Other): Women assigned to the control arm of the study received conventional prenatal and postpartum clinic care.
  Interventions: Other: Conventional prenatal/postpartum care

INTERVENTIONS:
Behavioral: Targeted Nurse Home Visits — Advanced practice nurses provide targeted behavioral interventions during home visits. These visits were in addition to regularly scheduled conventional prenatal and postpartum clinic care. Specific protocols guided nurse interventions related to tobacco use, substance use and misuse, stress management, dental health, maternal infections, perinatal depressive symptoms, family violence, reproductive life plans and continuity of care. Home visits were continued in the postpartum period (through 18 months post-delivery) with a continued focus on risk factors identified during the prenatal period and internatal health care.
  Arms: Targeted Nurse Home Visits
Other: Conventional prenatal/postpartum care — Women in this group received conventional prenatal care and postpartum clinic care.
  Other Names: standard medical prenatal and postpartum care

SUMMARY:
Women with a history of a prior preterm birth (PTB) have a high probability of a recurrent preterm birth. Some risk factors and health behaviors that contribute to PTB may be amenable to intervention. Home visitation is a promising method to deliver evidence based interventions. We evaluated a system of care designed to reduce preterm births and hospital length of stay in a sample of pregnant women with a history of a PTB. All participants (N = 211) received standard prenatal care. Intervention participants (N = 109) also received home visits by certified nurse-midwives guided by protocols for specific risk factors (e.g., depressive symptoms, abuse, smoking). Data was collected via multiple methods and sources including intervention fidelity assessments. Average age was 27.6 years. Racial breakdown mirrored local demographics. Most women had a partner, a high school education, and Medicaid. Enhanced prenatal care by nurse-midwife home visits may limit some risk factors and shorten intrapartum length of stay for women with a prior PTB. This study contributes to knowledge about evidence-based home visit interventions directed at risk factors associated with PTB.

DETAILED DESCRIPTION:
Preterm births (PTBs) are the leading cause of death in infants under the age of one. Tennessee (TN) is one of the lowest ranking states in the US for rates of PTBs (46th) and infant mortality (48th). Costs for neonatal care increase exponentially with decreasing gestational age, and there are lifelong consequences for families and communities. Despite medications and improved diagnostic tools, a 27% increase in PTBs has occurred in the past 20 years. With a history of one PTB, the probability of another PTB is approximately 30%. The risk of having another PTB rises to almost 70% if the woman has a history of more than one PTB. Relationships between a variety of factors (e.g., African American race, smoking, short interval between pregnancies, socio-environmental stressors) likely contribute to TN's high rate of PTBs. Several interventions have been identified to reduce PTBs and improve maternal and infant health indicators but with varying success; administering intramuscular injections of progesterone between 16 and 36 weeks gestation, providing some prenatal care in the home of women with a high risk pregnancy, increasing the interval between pregnancies, and reducing social factors that negatively impact health, such as smoking, substance abuse and stress.

The overall purpose of this study was to determine if a combined medical and biobehavioral intervention would prevent PTBs and reduce healthcare costs in a sample of women who have had a prior PTB. The medical intervention was conventional prenatal and postpartum clinic care. The biobehavioral intervention included certified nurse midwife home visitors who engaged women in an integrated System of Care (SOC) during their prenatal care. Care continued during the first 18 months of the infant's life by maternal-child nurse visitors. Home visits were in addition to regularly scheduled conventional prenatal and postpartum clinic care. Main study questions were:

Is there a difference in: 1) the length of gestational age of infants of high-risk pregnant women who receive the medical intervention and high-risk pregnant women who receive the SOC? 2) in health care costs between women who receive the medical intervention and the SOC? 3) intervals between the current pregnancy and a subsequent pregnancy across groups? and 4) in length of gestational age of current infant with gestational age of index prior preterm birth?

ELIGIBILITY:
Inclusion Criteria:

* Documented history of previous preterm delivery. Defined as delivery from 20 weeks to 36 weeks 6 days gestation.
* Proven pregnancy
* Reside in Davidson County, Tennessee (TN) or surrounding county in 90 mile driving radius.
* Less than 24 weeks gestation at enrollment
* Will receive prenatal care at a Vnderbilt University Medical Center (VUMC) clinic
* Willing to accept nurse home visits and be randomly assigned to conventional care or care with home visits
* Speaks and understands English
* Between the ages of 18 and 40 years.

Exclusion Criteria:

* Known fetal anomaly that can not be managed conservatively or fetal demise
* Maternal medical or obstetrical complications including:

  * Current or scheduled cervical cerclage
  * PROM in current pregnancy prior to enrollment
* Participation in an antenatal study in which the clinical status or intervention may influence gestational age at delivery
* Profound mental dysfunction or under guardianship

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 236 (Actual)
Dates: Start 2006-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Lutenbacher, PhD, Principal Investigator — Vanderbilt University; Patricia Temple, MD, MPH, Principal Investigator — Ohio State University and Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lutenbacher M, Gabbe PT, Karp SM, Dietrich MS, Narrigan D, Carpenter L, Walsh W. Does additional prenatal care in the home improve birth outcomes for women with a prior preterm delivery? A randomized clinical trial. Matern Child Health J. 2014 Jul;18(5):1142-54. doi: 10.1007/s10995-013-1344-4. PMID 23922160
- [Result] Karp SM, Howe-Heyman A, Dietrich MS, Lutenbacher M. Breastfeeding initiation in the context of a home intervention to promote better birth outcomes. Breastfeed Med. 2013 Aug;8(4):381-7. doi: 10.1089/bfm.2012.0151. Epub 2013 Mar 13. PMID 23484671

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The sample consisted of pregnant women receiving prenatal care with a (physician or nurse-midwife) at a large regional medical center in the Southeastern U.S. from April, 2007 through January, 2010.
Groups:
- Intervention Group: Advanced practice nurses provide targeted behavioral interventions during home visits. These visits were in addition to regularly scheduled conventional prenatal and postpartum clinic visits. Specific protocols guided nurse interventions related to tobacco use, substance use and misuse, stress management, dental health, maternal infections, perinatal depressive symptoms, family violence, reproductive life plans and continuity of care. Home visits were continued in the postpartum period (through 18 months post-delivery) with a continued focus on risk factors identified during the prenatal period and internatal health care.
- Control Group: Women assigned to the control arm of the study received conventional prenatal and postpartum clinic care.
  Conventional prenatal and postpartum clinic care : Women in this group received conventional prenatal care and postpartum clinic care.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 122 | 114
Completed | 109 | 102
Not Completed | 13 | 12
Not completed — Withdrawal by Subject | 3 | 1
Not completed — disenrolled due to pregnancy loss | 3 | 5
Not completed — found not to meet eligibility criteria | 3 | 4
Not completed — did not meet assignment criteria | 4 | 2

BASELINE CHARACTERISTICS:
Population: We analyzed data for participants who remained in the study for at least four weeks following enrollment. The final sample totaled 211 women: 109 intervention and 102 controls.
Groups:
- Treatment Group: Advanced practice nurses provide targeted behavioral interventions during home visits. These visits were in addition to regularly scheduled conventional prenatal and postpartum clinic visits. Specific protocols guided nurse interventions related to tobacco use, substance use and misuse, stress management, dental health, maternal infections, perinatal depressive symptoms, family violence, reproductive life plans and continuity of care. Home visits were continued in the postpartum period (18 months post-delivery) with a continued focus on risk factors identified during the prenatal period and internatal health care.
- Control Group: Women assigned to the control arm of the study received conventional prenatal and postpartum clinic care.
  Conventional prenatal and postpartum clinic care: Women in this group received conventional prenatal care and postpartum clinic care.
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 109 | 102 | 211
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 109 | 102 | 211
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.4 (5.5) | 27.8 (5.2) | 27.6 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 102 | 211
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 41 | 34 | 75
  White | 67 | 67 | 134
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 109 | 102 | 211
Marital Status [Number; unit: participants]
  Married or Partnered | 78 | 75 | 153
  Divorced or Separated | 4 | 8 | 12
  Never Married | 27 | 19 | 46
Type of insurance [Number; unit: participants]
  Medicaid | 64 | 62 | 126
  Private/Champus | 44 | 36 | 80
  None/self pay | 0 | 3 | 3
  Unknown or not reported | 1 | 1 | 2
Level of education in years [Mean (Standard Deviation); unit: years] | 13.2 (2.5) | 13.4 (2.6) | 13.3 (2.6)
Gestational age at enrollment in weeks [Mean (Standard Deviation); unit: weeks] | 15.43 (4.57) | 15.29 (4.57) | 15.43 (4.57)

OUTCOME MEASURES:

1. Primary Outcome: Infant Gestational Age
Description: Infant gestational age was determined by the weeks and days gestation documented in the maternal delivery record.
Time Frame: Time of delivery
Population: ITT analysis used with all participants that birth information could be obtained.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 108 | 102
weeks | 38.14 [36.57 to 39.29] | 38.14 [36.29 to 39.14]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; The original proposed sample size for this study was 300. This sample size was based on previous evidence that indicated that a reduction of 15% in the rate of preterm birth would be detectable with groups of 150. Because of concerns with systemic changes in the study's health care delivery environment, an interim analysis was conducted after 200 women had delivered. As a result of that analysis a decision was made to stop recruitment; Test type: Superiority or Other; p = .64, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Maternal Length of Stay at Delivery
Description: Number of maternal hospital days associated with delivery
Time Frame: Hospital discharge point following delivery
Population: Of the 211 participants, data on length of stay at delivery were available for 194 women. The most common reason for the lack of this information was that the birth did not take place at the study's medical center.
Measure: Median (Full Range); unit: days
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 101 | 93
days | 2 [1 to 12] | 3 [0 to 40]

ADVERSE EVENTS:
Arm/Group | Intervention Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/122 | 0/114
Other Adverse Events (participants affected / at risk) | 0/122 | 0/114

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No